CLINICAL TRIAL: NCT06557824
Title: Efficacy of Pulmonary Rehabilitation Combined With Speleotherapy in Children With Bronchial Asthma: a Retrospective Study.
Brief Title: Pulmonary Rehabilitation Combined With Speleotherapy in Children With Bronchial Asthma
Status: Completed | Type: Observational
Sponsor: University School of Physical Education, Krakow, Poland (Other)
Collaborators: Andrzej Frycz Modrzewski Krakow University (Other); Sanatorium Edel (Unknown); Health Resort "Wieliczka" Salt Mine (Unknown)
Responsible Party: Principal Investigator, Sylwia Mętel, PhD, MSc, working as Assistant Professor in Insitute of Applied Sciences, Faculty of Motor Rehabilitation, University of Physical Education in Krakow, University School of Physical Education, Krakow, Poland
Other Study IDs: AWF-EDEL 1/2024
Record Dates: First submitted 2024-07-13; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Asthma in Children
Keywords: asthma; children; subterranean therapy; 6MWT; exhaled nitric oxide
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: speleotherapeutic intervention — In the study, medical records of 415 Czech children diagnosed with bronchial asthma who took part in speleotherapeutic intervention between January 2022 and October 2023 were analysed.

SUMMARY:
The goal of this retrospective study is to learn about the effects of rehabilitation and treatment stays combined with speleotherapy in children with asthma. Medical records of 415 patients with this clinical diagnosis were analyzed and the main question was:

• Does speleotherapeutic intervention increase distance in 6-Minute Walk Test (6MWT) and influence spirometry parameters and fractional exhaled nitric oxide concentration (FeNO) in children with asthma?

DETAILED DESCRIPTION:
Background: Bronchial asthma is the leading cause of chronic disease and missed school days in children. The aim of the study was to evaluate pulmonary function and exercise tolerance in children with asthma who underwent speleotherapeutic intervention (STI) between January 2022 and October 2023 at Sanatorium Edel in Zlaté Hory.

Methods: Medical records of 415 patients with clinical diagnosis of bronchial asthma (J45.9, J45.0, J45, J45.8, J45.1) were analysed. The patients attended rehabilitation and treatment stays with a median length of 32 days combined with an average number of 15 speleotherapy sessions. The spirometry parameters, fractional exhaled nitric oxide concentration (FeNO), and 6-Minute Walk Test (6MWT) distance were measured before and after STI.

ELIGIBILITY:
Inclusion Criteria:

- Children with asthma who partcipated in speleotherapeutic intervention in Sanatorium Edel in Zlate Hory

Exclusion Criteria:

* Patients with incomplete data

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Medical records of 415 patients with clinical diagnosis of bronchial asthma (J45.9, J45.0, J45, J45.8, J45.1) were analysed.
Sampling Method: Non-Probability Sample
Enrollment: 415 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Forced expiratory flow in 1 second | January 2022 and October 2023
  Forced expiratory flow in 1 second, pp=percent predicted (FEV1 [pp]) to assess the pulmonary function in children with asthma before and after speleotherapeutic intervention.
6-Minute Walk Test (6MWT) | January 2022 and October 2023
  6-Minute Walk Test (6MWT) distance was measured to assess exercise tolerance in children with asthma before and after speleotherapeutic intervention.
Peak expiratory flow (PEFR [pp]) | January 2022 and October 2023
  Peak expiratory flow (PEFR [pp]) to assess the pulmonary function in children with asthma before and after speleotherapeutic intervention.

SECONDARY OUTCOMES:
Fractional exhaled nitric oxide concentration (FeNO) | January 2022 and October 2023
  The fractional exhaled nitric oxide concentration (FeNO) was measured to recognize the presence of eosinophillic inflammation involving the bronchial tree in children with asthma before and after speleotherapeutic intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sylwia Mętel, PhD, Principal Investigator — University of Physical Education in Krakow
Locations (1):
- University of Physical Education in Krakow, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No
Open access journals